CLINICAL TRIAL: NCT05213871
Title: Effect of Instrument-assisted Soft Tissue Mobilization Versus Myofascial Release in Treatment of Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Abdelfattah Hanafy shewail, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fatma_phd_2022
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Neck Pain; Soft Tissue Injuries
MeSH Terms: conditions — Neck Pain; Soft Tissue Injuries | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM group (Experimental): Group (A) will receive IASTM on the right upper trapezius and levator scapulae twice a week for four weeks in addition to a postural correction program.
  Interventions: Other: Instrument-assisted soft tissue mobilization; Other: Postural correction exercises (PCE)
- myofascial release group (Experimental): Group (B) will receive a myofascial release on the right upper trapezius and levator scapulae twice a week for four weeks in addition to the postural correction program.
  Interventions: Other: Myofascial release therapy; Other: Postural correction exercises (PCE)

INTERVENTIONS:
Other: Instrument-assisted soft tissue mobilization — For IASTM, the subject will be seated in a comfortable position. The subject's forehead will be rested on his/her forearm on a table in front of him/her. A lubricant (Vaseline) will be applied to the skin around the neck area prior to treatment and the M2T blade will be cleaned with an alcohol pad. The M2T blade will be used, at an angle of 45 without causing discomfort or pain, from the muscle origin to its insertion (sweeping technique), for approximately 3 min. Subjects will be instructed to put an ice pack on the area if they feel any burning sensations after the session. This procedure will be repeated twice a week for four weeks.
  Arms: IASTM group
Other: Myofascial release therapy — Firstly, the subject will lay supine with no pillow under his/ her head then the subject will rotate his/her head and neck away from the side which will be treated. Therapist will sit or stand at the corner, edge or top of the treatment table and therapist will place one hand proximal to the shoulder with skin on skin and therapist's fingers pointing towards the subject's elbow on the same side. Other hand of the therapist will be placed inferior to the subject's jaw (body of the mandible), using it as a handle, with fingers pointing towards the top of the subject's head. Then therapist will lean into the subject to the tissue depth barrier, wait and follow each subtle release three-dimensionally. Therapist should avoid forcing the tissue or slipping or gliding over the skin. The technique should be applied for at least five minutes for optimal results. This procedure will be repeated twice a week for four weeks.
  Arms: myofascial release group
Other: Postural correction exercises (PCE) — Postural correction exercises will be applied for patients in groups A and B. This program will be conducted according to the protocols of exercise will be performed as 3 sets of 10 repetitions each for 2 times/ week for 4 weeks. The patients will be instructed to continue the exercises as a daily home program to influence the self-correction kinesthetic awareness. Exercises will be performed while the patients in a neutral sitting posture

SUMMARY:
Mechanical neck pain has become a major health problem recently, affecting around one-year prevalence ranging from 42 to 67% in young adults aged 20-24 years causing pain and functional deficits. No study has been conducted before to investigate the effect of Instrument assisted soft tissue mobilization (IASTM) with mechanical neck pain on university students involved in distance learning.

DETAILED DESCRIPTION:
Mechanical neck pain is a major social and economic burden. It showed a one-year prevalence ranging from 42 to 67% in young adults aged 20-24 years. Treatment of neck pain is costly in terms of utilization of health care services, disability, compensation payments and lost work productivity. With the increasing prevalence of pain and disability associated with musculoskeletal impairments, it is essential to identify the most efficacious interventions to maximize patient outcomes and decrease the societal burden.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age will be between 18-25 years old.
2. Subjects with mechanical neck pain localized to cervical and periscapular region.
3. Subjects with at least one trigger point in the upper trapezius and/or levator scapulae muscles
4. Subjects should report mechanical neck pain of at least 30 mm on a visual analogue scale (VAS). The scale is ranged from 0 mm (no pain) to 100 mm (worst imaginable pain).
5. Subjects who use computers daily for at least two hours and are involved in distance learning for at least three months.

Exclusion Criteria:

1. Any specific neck pathology as radiculopathy, rheumatoid arthritis, and systemic diseases.
2. Sensory problems at mid or upper back
3. A tendency to hemorrhage or anticoagulation treatment. And nonsteroidal pain medication
4. History of head and upper trunk trauma or surgery.
5. Signs of severe pathology such as malignancy, fractures of the cervical spine, cervical radiculopathy or myelopathy, or vascular syndromes such as vertebrobasilar insufficiency.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessment | at baseline and after 4 weeks of intervention
  Assessing the change in pain intensity via using visual analogue scale which will be used to examine pain intensity. It consists of a continuous 10 cm line. The patient will be instructed to place a vertical mark on the line to indicate his/her pain, ranging from no pain or discomfort (0), to the worst pain he/she could possibly feel . Using the visual analogue scale allows the patient freedom to record and not restricting him by numbers.
Neck disability index | at baseline and after 4 weeks of intervention
  Assessing the change in neck disability via using Neck disability index which is is a self-reported outcome measure which is commonly used to determine the perceived disability in patients with neck pain. It consists of 10 items; 7 related to activities of daily living, (ADL), 2 related to pain, and 1 related to concentration. Each item is scored from 0-5 and the total score is expressed as percentage, with higher scores corresponding to greater disability.
Muscle pressure intensity | at baseline and after 4 weeks of intervention
  Assessing the change in Muscle pressure intensity via using Pressure Algometer which is a handheld device that applies a manual pressure stimulus to assess pressure intensity. It has been broadly used and validated. A pressure threshold algometer will be used to measure the pressure pain threshold of a Trigger points of the upper trapezius and levator scapulae muscle before and aftertreatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Hanafy, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Misr university for scientific and technology, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shewail F, Abdelmajeed S, Farouk M, Abdelmegeed M. Instrument-assisted soft tissue mobilization versus myofascial release therapy in treatment of chronic neck pain: a randomized clinical trial. BMC Musculoskelet Disord. 2023 Jun 3;24(1):457. doi: 10.1186/s12891-023-06540-5. PMID 37270471